CLINICAL TRIAL: NCT04090918
Title: Novel Methods for Characterizing Patients With Post-operative Atrial Fibrillation Secondary to Abdominal Surgery (A SECAFIB-SURG Sub-study)
Brief Title: Novel Methods for Characterizing Patients With Post-operative Atrial Fibrillation Secondary to Abdominal Surgery
Status: Withdrawn | Type: Observational
Why Stopped: It was not possible to ensure sufficient recruitment of patients to complete the study.
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Valdorff Madsen, Principal Investigator, Frederiksberg University Hospital
Other Study IDs: H-19033687
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Surgery--Complications
Keywords: post-operative atrial fibrillation; abdominal surgery; left atrial strain; atrial remodelling
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A venous blood sample (approximately 30 mL) and a urine sample (approximately 30 mL) will be collected for a Research biobank. Blood samples will be collected in EDTA- and serum tubes, respectively, extracting plasma (from the EDTA tube) and serum (from the serum tube). Samples are subsequently immediately frozen and transported on dry ice to a -80 degree freezer at Copenhagen University's Faculty of Health and Medical Sciences. Samples will be analysed when the last sample has been collected. Analyses will focus on markers of oxidative stress, coagulation abnormalities (factors II, VII, X and von Willebrand Factor) as well as fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Abdominal surgery with POAF: Twenty patients undergoing abdominal surgery with new-onset atrial fibrillation
  Interventions: Diagnostic Test: Cardiac examination programme 3 months after abdominal surgery
- Group 2: Abdominal surgery without POAF: Twenty patients undergoing abdominal surgery without new-onset atrial fibrillation matching patients in group 1 on age, sex and comorbidities.
  Interventions: Diagnostic Test: Cardiac examination programme 3 months after abdominal surgery

INTERVENTIONS:
Diagnostic Test: Cardiac examination programme 3 months after abdominal surgery — Blood- and urine sampling, electrocardiogram, wavECG (Myovista), transthoracic echocardiography, Finapres, cardiac magnetic resonance imaging

SUMMARY:
Purpose The primary purpose of the current project is to characterize unselected patients undergoing surgery developing post-operative atrial fibrillation (POAF), ultimately leading to a new risk-stratification model.

Background and rationale According to rather scarce existing reports, it is estimated that 10% will develop POAF following abdominal surgery. It remains a challenge for the clinicians to predict which patients are at risk. POAF can be difficult to diagnose, as symptoms are often vague. Hence, the diagnosis may remain underreported leaving many patients without adequate treatment. Untreated atrial fibrillation is associated with increased morbidity and mortality, especially due to an increased risk of ischemic stroke.

Methods Three-hundred adult patients admitted for surgery at the Digestive Disease Center at Bispebjerg Hospital will be examined by heart rhythm monitoring during hospitalization, i.e. pre-, peri- and postoperatively in the main SECAFIB-SURG study. Twenty study participants who develop POAF and 20 without POAF matched with these on sex, age and co-morbidity, will undergo additional cardiovascular examinations three months after surgery in the current sub-study. All patients will be followed for at least one year after surgery. The study is scheduled for completion within two years, commencing in January 2020.

Perspective Creating a POAF risk-stratification model for patients undergoing abdominal surgery, could ensure timely diagnosis and treatment, hence, preventing complications associated with POAF.

DETAILED DESCRIPTION:
Background and rationale Post-operative AF (POAF) appears to be common in relation to abdominal surgery affecting between 8% and 18%, however the incidence is not well reported,1 and the SECAFIB-SURG study aims at reporting this.

A number of risk-stratification models exist in the general population and in cardiac surgery patients, but it remains challenging to predict which patients will develop POAF in non-cardiac surgery patients.2-5 Diagnosing POAF is important, as recent data from the Framingham population suggest that secondary AF (AF occurring during a concomitant medical condition, e.g. surgery) is not a benign condition.6,7 Studies have found an association between POAF in relation to non-cardiac surgery and increased risk of post-operative mortality and stroke.8-10 Despite this, the current perception is that POAF is self-limiting and merely a result of the physiological stresses of surgery, why continuous anti-coagulation and referral for a cardiologist is not necessarily recommended.11-13 Well-known factors associated with AF in the general population is age, hypertension, heart failure, myocardial infarction, heart valve disease and diabetes.14 In general surgery important risk factors of AF is age (age 65-74, OR 2.08; age >85, OR 3.56), hypertension (OR 3.66), heart failure (OR 1.64), thyroid disease (OR 6.29), laparotomy (vs laparoscopy, OR 3.30) and duration of surgery (> 600 min, OR 1.38).1 The pathophysiology of AF is however incompletely comprehended.14-16 Structural remodelling of the atria and electrical pathways, oxidative stress, inflammation, calcium overload, myofibroblast activation and microRNAs are suspected implicated in AF initiation and progression.14-17 Improved understanding of the pathophysiology of AF and improved diagnostic tools for predicting POAF is needed. In the current study, blood samples will focus on markers of cardiac surcharge (troponins and natriuretic peptide)18,19, inflammation20-22 and microRNAs associated with AF.23-25 Urine samples will focus on oxidative stress markers.22,26,27 Electrocardiogram (ECG) will focus on short and prolonged p-wave, and p-wave terminal force in lead V1 (PTFV1) which are correlated with AF.28 Myovista (HeartSciences, Southlake, Texas, USA) a novel type of ECG (wavECG) utilizing continues wavelet transform signal processing, appears to identify left ventricular diastolic dysfunction (LVDD),29 which is associated with AF in other studies.16,30-32 Finapres Nova (Enschede, The Netherlands) is a continuous blood pressure monitor which will be used for non-invasive hemodynamic monitoring, e.g. beat-to-beat cardiac output, stroke volume, cardiac contractility, left ventricular ejection time and total peripheral resistance.33 Oral glucose tolerance test performed during monitoring with Finapres might demask peripheral vascular dysfunction.34 Speckle-tracking and strain analysis of the left atrium (LA) by transthoracic echocardiography (TTE) is in some studies able improve AF risk-prediction.35-39 Cardiac magnetic resonance imaging (CMRI) with late gadolinium enhancement (LGE) has been used to quantify atrial structural remodelling, fibrosis and function, and has been used to improve prediction of favourable outcome of patients undergoing ablation for AF.40-43

Purpose The study aims at characterizing patients developing POAF by novel methods to improve risk stratification of patients undergoing abdominal surgery.

Methods Prospective, single-centre, case-control study of patients undergoing abdominal surgery.

The current study is a sub-study of SECAFIB-SURG. Study participants will be identified among those enrolled in the SECAFIB-SURG study (study ID: 68605) who have agreed to be contacted if they developed POAF or matched on age and gender with someone who did. POAF is defined as new-onset AF developing from surgery until discharge and diagnosed by specialists in Cardiology or Anaesthesiology on ECG or heart rhythm monitoring for at least 30 seconds duration or three recurrent episodes of AF. The Investigator (Department of Cardiology at Bispebjerg-Frederiksberg Hospital) will ensure signed informed consent.

Statistical considerations LA strain analysis has not been performed in this patient group. LA strain has predicted recurrence of AF in patients who have undergone radiofrequency ablation.23,24 In one study, patients with recurrent AF had LA strain mean of 18.4% while those without recurrence had a LA strain mean of 25.5%23. In another study, patients with recurrent AF had LA strain mean of 9.7% while those without recurrence had a LA strain mean of 16.2%.24 With 95% power and alpha 0.05, and enrolment ratio 1:1, 5 patients with - and 5 patients without - are required to identify significant difference in LA strain mean between the two groups. The current population is however expected more heterogenous that those undergoing radiofrequency ablation and as the study is explorative it will include 20 patients with POAF and 20 matched controls without POAF. Follow-up will remain unchanged from the main study, i.e. one year from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the SECAFIB-surg study
* Signed informed consent

Exclusion Criteria:

* Ongoing inflammation or infection
* Connective tissue disease
* Active cancer diagnosis
* Follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, single-centre, case-control study of patients undergoing abdominal surgery.
  The current study is a sub-study of SECAFIB-SURG. Study participants will be identified among those enrolled in the SECAFIB-SURG study (H-19033464) who have agreed to be contacted if they developed POAF or matched on age and gender with someone who did.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal left atrial strain | Three months after abdominal surgery
  Left atrial strain abnormality as measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Number of patients with clinical events after surgery | From surgery until 1 year after surgery
  Clinical events defined as: reoperation; occurrence/recurrence of AF; ischemic stroke or transient ischemic attack; all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer V Madsen, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No data has been obtained.